CLINICAL TRIAL: NCT06294444
Title: Effects of CIMT With and Without Mirror Therapy on Upper Limb Function in Children With Hemiplegic Cerebral Palsy
Brief Title: Comparison of Constraint Induced Movement Therapy and Mirror Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REC/RCR&AHS/23/0741
Record Dates: First submitted 2023-12-26; First posted 2024-03-05 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: mCIMT, Hemiplegia, Mirror therapy
MeSH Terms: conditions — Hemiplegia | interventions — Constraint Induced Movement Therapy; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: Participants will get separate treatment protocol and possible efforts will be put to mask the both groups about their treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint induced Movement Therapy (Experimental): Group of 15 members will be given constraint induced movement therapy for 6 weeks.
  Interventions: Other: Constraint Induced Movement Therapy
- Mirror therapy group (Experimental): Group of 15 members will be given modified constraint induced movement therapy with mirror theray for 6 weeks.
  Interventions: Other: Mirror therapy

INTERVENTIONS:
Other: Constraint Induced Movement Therapy — Group A: This group patients will be treated with mCIMT, the forced use of the affected arm by restraining the unaffected arm, with a sling or a hand splint, during dedicated exercise sections or usual ADLs (90% of waking hours).Massed practice (eight hours of exercise) of the affected arm through a shaping method, where shaping involves a commonly operant conditioning method in which a behavioural objective (in this case 'movement') is approached in small steps of progressively increasing difficulty. The participant is rewarded with enthusiastic approval for improvement, but never blamed or punished for failure. This therapy will be given 4hrs daily for 6 weeks. The results will be based upon pre and post evaluation.
  Other Names: Mirror Therapy
  Arms: Constraint induced Movement Therapy
Other: Mirror therapy — Group B: These patients will be treated with mCIMT and mirror therapy. Children were taught repetitive symmetrical upper limbs exercises: with modelling-clay in each hand to elicit bilateral thumb-finger pinch and grasping. They performed these during a 15-minute daily routine at home with mCIMT (forced use of arm and massed practice 4hrs of exercise of affected arm). This combination of therapy will be given for 6 weeks. The results will be seen through pre and post evaluation.
  Arms: Mirror therapy group

SUMMARY:
Hemiplegia in infants and children is a type of Cerebral Palsy that results from damage to the part (hemisphere) of the brain that controls muscle movements. This damage may occur before, during or shortly after birth. The term hemiplegia means that the paralysis is on one vertical half of the body. The aim of this study will be the to know the effect of mCIMT with and without mirror therapy on upper limb function in children with hemiplegic cerebral palsy. A randomized control trial will be conducted at Sheikh Zayed Hospital, RYK through convenience sampling technique on 30 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and group B. Group A will be treated with mCIMT and Group B will be treated with mCIMT and mirror therapy. Outcome measure will be conducted through pain and disability questionnaire after 6 weeks. Data will be analyzed using SPSS software version 21. After assessing normality of data by Shapiro - wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups. mCIMT with and without mirror therapy will be applied in patients with hemiplegic cerebral palsy to see the effect on upper limb function.

DETAILED DESCRIPTION:
Patients who will meet the inclusion criteria will be recruited by convenience sampling technique and allocated to groups by simple randomization process by sealed opaque enveloped labeled as 0 for Group A and 1 for Group B.

After taking consent from the patients parents with hemiplegic CP of both genders will be randomized into two equal groups. Patients from physical therapy department will be assessed with CHEQ and Melbourne Assessment of the Unilateral Upper Limb Function (MAULF) and the Functional Hand Grip Test (FHGT) . At start of study, a formal educational session, lasting about 30 min will be given by physiotherapist.

Group A: This group patients will be treated with mCIMT, the forced use of the affected arm by restraining the unaffected arm, with a sling or a hand splint, during dedicated exercise sections or usual ADLs (90% of waking hours).Massed practice (eight hours of exercise) of the affected arm through a shaping method, where shaping involves a commonly operant conditioning method in which a behavioural objective (in this case 'movement') is approached in small steps of progressively increasing difficulty. The participant is rewarded with enthusiastic approval for improvement, but never blamed or punished for failure. This therapy will be given 4hrs daily for 6 weeks. The results will be based upon pre and post evaluation.

Group B: These patients will be treated with mCIMT and mirror therapy. Children were taught repetitive symmetrical upper limbs exercises: with modelling-clay in each hand to elicit bilateral thumb-finger pinch and grasping. They performed these during a 15-minute daily routine at home with mCIMT (forced use of arm and massed practice 4hrs of exercise of affected arm). This combination of therapy will be given for 6 weeks. The results will be seen through pre and post evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Medically diagnosed with Hemiplegic CP
* Age ranges btween3-12 years
* Hemiplegic CP with motor disability
* No major contractures of upper limb muscle
* Both genders were included
* Able to follow command
* No orthopedic surgery during the previous six months(8)

Exclusion Criteria:

* Functional limb
* Patients with contracture
* Patient with sensory,cognitive and perceptual disorders
* Patient with seizures
* Patient with orthopedic surgery

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
fine motor skills | 6weeks
  The Melbourne Assessment 2 (MA2): a test of quality of unilateral upper limb function. Is a criterion-referenced test for children aged 2.5 to 15 years with neurological impairments providing measurement of four elements of upper limb movement quality: range of movement, accuracy, dexterity and fluency.
  FHGT: The subject holds the dynamometer in the hand to be tested, with the arm at right angles and the elbow by the side of the body. The handle of the dynamometer is adjusted if required - the base should rest on the first metacarpal (heel of palm), while the handle should rest on middle of the four fingers. When ready the subject squeezes the dynamometer with maximum isometric effort, which is maintained for about 5 seconds. No other body movement is allowed. The subject should be strongly encouraged to give a maximum effort.
  MMT: Manual Muscle Testing Grades 0-5

CONTACTS AND LOCATIONS:
Overall Officials: Hurriya Sehar, MS*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Imran Amjad, Lahore, Punjab Province
  - Riphah International University, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oliva-Sierra M, Rios-Leon M, Abuin-Porras V, Martin-Casas P. [Effectiveness of mirror therapy and action observation therapy in infantile cerebral palsy: a systematic review]. An Sist Sanit Navar. 2022 Aug 16;45(2):e1003. doi: 10.23938/ASSN.1003. Spanish. PMID 35972309